CLINICAL TRIAL: NCT07168863
Title: Incidence and Risk Factors of Acute Pancreatitis Following EUS-Guided Fine Needle Biopsy (EUS-FNB)
Brief Title: EUS-guided FNB-induced PANCREatitis Assessment
Acronym: EUS-PANCREA
Status: Recruiting | Type: Observational
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, Mehdi Mohamadnejad, Associate Professor of Medicine, University of Tehran
Other Study IDs: IR.TUMS.DDRI.REC.1404.010
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pancreatitis, Acute; EUS Guided Biopsy
Keywords: acute pancreatitis; EUS-guided FNB
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EUS-guided FNB — EUS-guided FNB from the lesions in the pancreatobiliary tract

SUMMARY:
This is a descriptive analytical study to investigate the prevalence and risk factors for pancreatitis after Endoscopic Ultrasonography-guided Fine Needle Biopsy (EUS-FNB) in patients at Shariati Hospital in Tehran. The study aims to identify risk factors for post-FNB pancreatitis to improve clinical protocols, reduce complications and treatment costs, and increase diagnostic accuracy for pancreatic and biliary tract diseases. The study will collect demographic and clinical data from all eligible patients undergoing EUS-guided FNB during the study period. Amylase and lipase levels will be measured in all enrolled patients 24 hours post-procedure. Pancreatitis will be diagnosed based on abdominal pain and amylase or lipase levels exceeding three times the normal range 24 hours after the procedure. The outcomes will be independently adjudicated by an expert gastroenterologist not involved in the EUS procedures by reviewing participants' medical records. The consensus definition will be applied as a diagnostic framework (rather than a strict definition) so that the adjudicator can use their best judgment in cases that does not strictly satisfy the criteria. The patients will be contacted 24-72 h after the procedure to follow-up on any potential complications. The study plans to enroll at least 300 patients.

DETAILED DESCRIPTION:
EUS-guided tissue acquisition is an advanced diagnostic procedure for evaluating and diagnosing pancreatic, ampullary, and biliary tract tumors due to its high accuracy and minimally invasive nature. However, a potential complication is acute pancreatitis. This can lead to serious clinical problems, including severe abdominal pain, prolonged hospitalization, and, in rare cases, life-threatening complications. EUS-guided FNA of pancreatic masses is infrequently associated with acute pancreatitis. The incidence of pancreatitis after FNA of solid and cystic pancreatic lesions is reported to be 0.64%, and 1.4%, respectively (1, 2). The designs of the tips of FNA and FNB needles are different, and it may have impact on the risk of pancreatitis after FNB. Personal observations of the researchers of this study suggest that the risk of pancreatitis is likely higher after EUS-FNB than EUS-FNA, however, the incidence of pancreatitis after EUS-guided FNB is not systematically studied. The purpose of this study is to determine the incidence of acute pancreatitis after EUS-FNB and identify the risk factors associated with post-EUS-FNB pancreatitis to help prevent and manage this complication, improve clinical outcomes, reduce treatment costs, and enhance diagnostic accuracy for pancreatic and biliary tract diseases. The study is a descriptive analytical study that will be conducted on patients referred to the endoscopy department of Shariati Hospital in Tehran who will undergo EUS-guided FNB.

Patient information, including demographic data and clinical characteristics, will be collected using specialized checklists based on clinical interviews, patient examinations, and review of patient records. The data collected will include gender, age, indication for FNB, history of acute or chronic pancreatitis, and technical details of the procedure, such as the needle brand and size, anatomical location of the biopsy, amount of normal pancreatic tissue the needle passes through, number of passes, and the biopsy site (stomach or duodenum).

All patients meeting the inclusion criteria will be enrolled in the study. Amylase and lipase levels will be measured in all enrolled patients 24 hours post-procedure. Pancreatitis will be diagnosed based on abdominal pain and amylase or lipase levels exceeding three times the normal range 24 hours after the procedure. The outcomes will be independently adjudicated by an expert gastroenterologist not involved in the EUS procedures by reviewing participants' medical records. The consensus definition will be applied as a diagnostic framework (rather than a strict definition) so that the adjudicator can use their best judgment in cases that does not strictly satisfy the criteria. The patients will be contacted 24-72 h after the procedure to follow-up on any potential complications. Patients who develop pancreatitis will receive standard diagnostic and therapeutic follow-up. The study plans to enroll at least 300 patients.

ELIGIBILITY:
Inclusion Criteria:

Inpatients and outpatients aged 18 years or older undergoing EUS-guided FNB from a solid or cystic lesion in one of the following locations:

* Pancreas
* Ampulla of Vater
* Distal CBD, defined as the intrapancreatic portion of the CBD where the FNB needle passes through the pancreas during biopsy

Exclusion Criteria:

* Patients who undergo concurrent ERCP in the same day
* Patients experiencing an ongoing episode of acute pancreatitis during EUS-FNB
* Patients undergoing EUS-guided FNA
* Uncorrectable coagulopathy (INR > 1.5)
* Uncorrectable thrombocytopenia (platelet < 50,000)
* Decline to participate in the study and sign the informed consent form
* Patients undergoing EUS-guided FNB from the proximal CBD where the FNB needle does not traverse the pancreas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive inpatients and outpatients aged 18 years or older undergoing EUS-guided FNB at Shariati Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-02-12 (Estimated); Study Completion 2027-03-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-EUS-FNB acute pancreatitis | From enrollment to three days after EUS-FNB
  Determining the incidence of acute pancreatitis after EUS-guided FNB from the pancreatobiliary lesions

SECONDARY OUTCOMES:
Factors associated with post-EUS-FNB pancreatitis | From enrollment to three days after EUS-FNB
  The secondary objectives are to determine the role of the following factors in the development of pancreatitis after EUS-guided FNB:
  * Gender
  * Age
  * Biopsy site
  * Dilation of the main pancreatic duct (PD) and common bile duct (CBD)
  * The amount of normal pancreatic tissue the needle passes through
  * Number of needle passes
  * Number of back and forth movement of the needle in each pass
  * Biopsy approach (transgastric or transduodenal)
  * History of pancreatitis
  * Type of lesion (solid vs. cystic)
  * Needle size
Incidence of moderate to severe post-FNB pancreatitis | From enrollment to one week after EUS-FNB
  The incidence of moderate to severe post-FNB pancreatitis will be assessed using Atlanta classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Shariati Hospital, Digestive Diseases Research Institute, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared for collaborative research after reviewing the requester's research protocol
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: IPD will be accessible following the study's publication and will remain available for three years.
Access Criteria: IPD will be shared for collaborative research after reviewing the requester's research protocol

REFERENCES:
- [Background] Eloubeidi MA, Gress FG, Savides TJ, Wiersema MJ, Kochman ML, Ahmad NA, Ginsberg GG, Erickson RA, Dewitt J, Van Dam J, Nickl NJ, Levy MJ, Clain JE, Chak A, Sivak MV Jr, Wong R, Isenberg G, Scheiman JM, Bounds B, Kimmey MB, Saunders MD, Chang KJ, Sharma A, Nguyen P, Lee JG, Edmundowicz SA, Early D, Azar R, Etemad B, Chen YK, Waxman I, Shami V, Catalano MF, Wilcox CM. Acute pancreatitis after EUS-guided FNA of solid pancreatic masses: a pooled analysis from EUS centers in the United States. Gastrointest Endosc. 2004 Sep;60(3):385-9. doi: 10.1016/s0016-5107(04)01714-6. PMID 15332028
- [Background] Magahis PT, Chhoda A, Berzin TM, Farrell JJ, Wright DN, Rizvi A, Hanscom M, Carr-Locke DL, Sampath K, Sharaiha RZ, Mahadev S. Risk of Pancreatitis After Endoscopic Ultrasound-Guided Fine-Needle Aspiration of Pancreatic Cystic Lesions: A Systematic Review and Meta-Analysis. Am J Gastroenterol. 2024 Nov 1;119(11):2174-2186. doi: 10.14309/ajg.0000000000002942. Epub 2024 Jul 5. PMID 38976379